CLINICAL TRIAL: NCT05830760
Title: Expression of Sodium Glucose Co-transporter2 in Myocardium From Patients With Aortic Valve Stenosis and With/Without Diastolic Heart Failure
Brief Title: Expression of Sodium-glucose Co-transporter 2 in Human Heart
Acronym: SGLT2-MICRA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: authorization obsolete
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8774
Record Dates: First submitted 2023-03-24; First posted 2023-04-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis
Keywords: human heart; myocardium; aortic valve stenosis; heart failure; sodium glucose cotransporter 2
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with aortic valve stenosis with heart failure (Experimental)
  Interventions: Biological: Myocardium biopsy
- patients with aortic valve stenosis without heart failure (Experimental)
  Interventions: Biological: Myocardium biopsy

INTERVENTIONS:
Biological: Myocardium biopsy — The expression of SGLT2 on small myocardium specimens harvested during aortic valve replacement operation in patients with aortic stenosis

SUMMARY:
The aim of the study is to evaluate the expression of Sodium Glucose Co-transporter 2 (SGLT2) in myocardium from patients with aortic stenosis. 2 groups of patients will be defined: Group A with diastolic heart failure and Group B without heart failure. The expression of SGLT2 will be measured on small myocardium specimens harvested during aortic valve replacement operation. This study should allow us to better understand the effect of glifozines in human heart failure.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years-old
* Patient with surgical aortic valve stenosis, with or without heart failure, in two equal-sized groups (40 subjects in each group)
* Subjects affiliated with a social security health insurance plan
* Subject able to understand the objectives and risks of the research and to give dated and signed informed consent

Exclusion Criteria:

* Infective endocarditis in aortic stenosis
* Severe coronary pathology associated with aortic stenosis
* Impossible to give the subject informed information (subject in emergency situation, difficulties in understanding the subject, ...)
* Subject under legal protection
* Subject under guardianship or curatorship
* Pregnancy and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To study the expression levels of SGLT2 in the myocardium of patients with surgical aortic stenosis | Day 0
  Measure of SGLT2 expression level by RT-PCR and
To study the SGLT2 tissue localization in the myocardium of patients with surgical aortic stenosis | Day 0
  SGLT2 expression level by immunofluorescence labeling

SECONDARY OUTCOMES:
Comparison of SGLT2 expression levels between heart failure and non-heart failure patients. | Day 0
  SGLT2 expression levels between the 2 groups of patients
Assess oxidative stress | Day 0
  Pro-oxidant response (fluorescence level of the redox-sensitive fluorescent probe DHE)
Evaluate the pro-inflammatory response by analysing the expression level of tissue activation molecules VCAM-1, ICAM-1, MCP-1 | Day 0
  Pro-inflammatory response: (VCAM-1, ICAM-1, MCP-1). Expression level of tissue activation molecules VCAM-1, ICAM-1, MCP-1 by RT-PCR, Western blot analysis and immunofluorescence labeling
Evaluate the pro-fibrotic response | Day 0
  Pro-fibrotic response: TGF beta, Ang II, AT1R, ACE, collagen; MMP-2, MMP-9. Expression level of molecules involved in tissue remodeling TGF beta, Ang II, AT1R, ACE, collagen, MMP-2, MMP-9 by RT-PCR, Western blot analysis and immunofluorescence labeling
Evaluate the pro-senescent response | Day 0
  Pro-senescent response: SA-beta-galactosidase activity, p53, p21, P16. Determination of senescence-associated beta-galactosidase activity on cardiac muscle cryosections, and expression level of senescence mediators p53, p21, p16 by RT-PCR, Western blot analysis and immunofluorescence labeling
Evaluate the pro-thrombotic response | Day 0
  Pro-thrombotic response: tissue factor. Expression level of coagulation cascade activator, tissue factor by RT-PCR, Western blot analysis and immunofluorescence labeling
Evaluate endothelial dysfunction | Day 0
  Endothelial response: eNOS, NO, nitrotyrosine. Expression level of eNOS and nitrotyrosine by RT-PCR, Western blot analysis and immunofluorescence labeling and NO formation using the NO-sensitive fluorescent probe, DAF-FM on heart muscle cryosections

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France